CLINICAL TRIAL: NCT03445975
Title: Preventing Pressure Ulcers (PU) in Intensive Care Units - The Effectiveness of Dry Washcloths Versus Usual Care: A Cluster-crossover Protocol
Brief Title: Washcloths Effectiveness in Preventing Pressure Ulcers
Acronym: Bathing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale San Donato (Other)
Responsible Party: Principal Investigator, Rosario Caruso, Head of Health Professions Research and Development Unit, Ospedale San Donato
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 84/INT/2016
Record Dates: First submitted 2018-02-15; First posted 2018-02-26 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Pressure Ulcer; Skin Ulcer
MeSH Terms: conditions — Pressure Ulcer; Skin Ulcer

STUDY DESIGN:
Intervention Model Description: This study had a cluster-crossover design, where each of the two involved ICUs was the cluster. The genaral aim was to test the effectiveness of a 3-in-1 perineal care washcloth versus standard of care (e.g., water and pH neutral soap) to prevent and treat pressure ulcers in ICUs. The study has been articulated in two phases, lasted three months each. In the first phase, from the 1st of February to the 2nd of May, the 3-in-1 perineal care washcloth procedure has been adopted by the ICU of San Donato Hospital (Milan, Italy), while the Cardiovascular Intensive Care Unit (CVICU) continued to adopt the standard procedure (water and pH neutral soap). In the second phase, from the 2nd of May to 31st of July, the two procedures have been switched between the two wards.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The 3-in-1 perineal care washcloth procedure has been adopted to deliver hygiene care (total or perineal) or baths
  Interventions: Procedure: 3-in-1 perineal care washcloths
- standard (No Intervention): The deliver of hygiene care (total or perineal) or baths has been performed using water and pH neutral soap

INTERVENTIONS:
Procedure: 3-in-1 perineal care washcloths — The 3-in-1 washcloth was used for daily routine perineal skin hygiene and after each diaper/underpad change. This procedure was intended for cleansing, moisturizing, and application of a barrier protection (dimeticone 3%). 3-in1 washcloths pH range is 3.5 to 5.0.
  Arms: Experimental

SUMMARY:
A monocentric cluster-crossover design has been used in this study to test the effectiveness of a 3-in-1 perineal care washcloth versus standard of care (e.g., water and pH neutral soap) to prevent and treat pressure ulcers in ICUs.

DETAILED DESCRIPTION:
This study had a cluster-crossover design, where each of the two involved ICUs was the cluster. The genaral aim was to test the effectiveness of a 3-in-1 perineal care washcloth versus standard of care (e.g., water and pH neutral soap) to prevent and treat pressure ulcers in ICUs. The study has been articulated in two phases, lasted three months each. In the first phase, from the 1st of February to the 2nd of May, the 3-in-1 perineal care washcloth procedure has been adopted by the ICU of San Donato Hospital (Milan, Italy), while the Cardiovascular Intensive Care Unit (CVICU) continued to adopt the standard procedure (water and pH neutral soap). In the second phase, from the 2nd of May to 31st of July, the two procedures have been switched between the two wards.

Adult patients (aged over 18 years old) requiring personal hygiene care (total or perineal) in ICU and CVICU of San Donato Hospital have been enrolled. Patients who present allergic reactions or sensitivity to the experimental procedure have been excluded. All the longitudinal data related to the presence/grading of pressure ulcer (PU) at every hygiene care (total or perineal) performed on the patients in ICU and CVICU have been collected.

The primary endpoint of the study is represented by PU during the hospitalization in ICUs, whis is expected to be reduced from 10% in the experimental clusters. A sample size composed by 240 patients (120 patients/group) has been calculated, following methodological approach for difference between proportions. The sample size was calculated to be representative in observing a 10% decrease in the onset of PU, with a 80% power and an alpha error equal to 0.05. This approach led to the detection of a clinical relevant difference to compare the effectiveness between the two different procedures.

Data collected for the study were recorded on data-collection sheets in hard copy format. Data were also collected after every hygiene procedure on patient-related characteristics, skin condition and general clinical status.

The comparison between the two clusters (i.e. ICU and CVICU) will be performed using Student's t-test for the continuous variables and the χ2 for the categorical ones. Treatment effectiveness will be evaluated through the difference between proportions of IAD and PU in Period 1 and Period 2. A decrease in the onset of IAD and PU is expected as the main endpoint, considering a 95% confidence interval. The data will be compared using generalized estimating equation (GEE). The variables that might have an influence on the prevalence/incidence measures (i.e., patient's characteristics and ICUs management/staffing) will be monitored. The Period will be considered a "within" factor and the procedure/cluster a "between" factor. The α significance level will be preventively set at 5%.

Data have been stored to a master file on the San Donato Hospital server. This is password-protected and only available to the Principal Investigator user. On completion of the project, identifying data have been removed from all the record.

ELIGIBILITY:
Inclusion Criteria:

* All patients (real-world)

Exclusion Criteria:

* Under 18 yo
* Patients who present allergic reactions or sensitivity to the experimental procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Pressure Ulcer | 6 months
  To describe the impact of 3-in-1 washcloths on pressure ulcers. Pressure ulcers are assessed using the classification proposed by the US-National Pressure Ulcer Advisory Panel (NPUAP)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, MI - Milano, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Beeckman D, Verhaeghe S, Defloor T, Schoonhoven L, Vanderwee K. A 3-in-1 perineal care washcloth impregnated with dimethicone 3% versus water and pH neutral soap to prevent and treat incontinence-associated dermatitis: a randomized, controlled clinical trial. J Wound Ostomy Continence Nurs. 2011 Nov-Dec;38(6):627-34. doi: 10.1097/WON.0b013e31822efe52. PMID 21952346
- [Background] Bliss DZ, Zehrer C, Savik K, Smith G, Hedblom E. An economic evaluation of four skin damage prevention regimens in nursing home residents with incontinence: economics of skin damage prevention. J Wound Ostomy Continence Nurs. 2007 Mar-Apr;34(2):143-52; discussion 152. doi: 10.1097/01.WON.0000264825.03485.40. PMID 17413828
- [Background] Truong B, Grigson E, Patel M, Liu X. Pressure Ulcer Prevention in the Hospital Setting Using Silicone Foam Dressings. Cureus. 2016 Aug 8;8(8):e730. doi: 10.7759/cureus.730. PMID 27630803
- [Background] Harris PN, Le BD, Tambyah P, Hsu LY, Pada S, Archuleta S, Salmon S, Mukhopadhyay A, Dillon J, Ware R, Fisher DA. Antiseptic Body Washes for Reducing the Transmission of Methicillin-Resistant Staphylococcus aureus: A Cluster Crossover Study. Open Forum Infect Dis. 2015 May 22;2(2):ofv051. doi: 10.1093/ofid/ofv051. eCollection 2015 Apr. PMID 26125031